CLINICAL TRIAL: NCT01785524
Title: Dietary Nitrate to Augment Exercise Training Benefits in Subjects With Type II Diabetes (DM) and Peripheral Arterial Disease (PAD)
Brief Title: Dietary Nitrate and Exercise to Augment Exercise Training Benefits in Subjects With DM+PAD
Acronym: DM+PAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jason Allen, Ph.D., Assistant Professor Doctor of Physical Therapy Program & Division of Cardiovascular Medicine, Duke University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00039608; 5R21HL113717-02 (NIH)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Peripheral Arterial Disease; Type II Diabetes Mellitus
Keywords: Cardiovascular Diseases; Vascular Diseases; Arterial Occlusive Diseases; Diabetes; Exercise; Functional Capacity
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Vascular Diseases; Arterial Occlusive Diseases; Diabetes Mellitus; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BR Juice (Beet-It Stamina Shot) & Supervised Exercise Training (Experimental): Subjects consume 70 ml of Beetroot Juice (Beet-It Stamina Shot) to assess acute effects of beverage supplementation at the start (between Testing Visits 1 & 2) and at the end of the trial (between Visits 3 & 4). It also allows for comparisons of the combination of beetroot juice and chronic training effects (between Visits 2 & 3) to when the subject has not consumed the beverage (Visits 1 & 4). All subjects will consume Beet-It Stamina Shot 3 hours prior to all beverage tolerance visits, Testing Visits 2 & 3 and for all supervised exercise training visits during the 12 week intervention.
  Interventions: Drug: Beetroot Juice (Beet-It Stamina Shot) and Exercise Training
- BR Juice Placebo and Exercise Training (Placebo Comparator): Subjects consume 70 ml of Beetroot Juice (Beet-It Stamina Shot; Placebo) to assess acute effects of beverage supplementation at the start (between Testing Visits 1 & 2) and at the end of the trial (between Visits 3 & 4). It also allows for comparisons of the combination of placebo beverage and chronic training effects (between Visits 2 & 3) to when the subject has not consumed the beverage (Visits 1 & 4). All subjects will consume Beet-It Stamina Shot (Placebo) 3 hours prior to all beverage tolerance visits, Testing Visits 2 & 3 and for all supervised exercise training visits during the 12 week intervention.
  Interventions: Other: Placebo Comparator Beverage (Beet-It Stamina Shot) & Exercise Training

INTERVENTIONS:
Drug: Beetroot Juice (Beet-It Stamina Shot) and Exercise Training — The beverage is high in inorganic nitrate and bottled and supplied by James White Drinks. This supplement will be used in conjunction with supervised exercise training.
  Other Names: James White Drinks
  Arms: BR Juice (Beet-It Stamina Shot) & Supervised Exercise Training
Other: Placebo Comparator Beverage (Beet-It Stamina Shot) & Exercise Training — The beverage is identical in look and taste to Beet-It Stamina Shot but with active ingredient removed. It is also bottled and supplied by James White Drinks. This placebo supplement will be used in conjunction with supervised exercise training.
  Other Names: James White Drinks
  Arms: BR Juice Placebo and Exercise Training

SUMMARY:
The hypothesis of this proposal is that in subjects with Type II diabetes mellitus (T2D) and peripheral arterial disease (PAD) with intermittent claudication (IC), regular consumption of a high nitrate supplement which raises plasma nitrite, in conjunction with 12 weeks of supervised exercise training at the limb ischemic threshold (SET) will produce a greater clinical benefit (increases in claudication onset time [COT] and peak walking time [PWT] relative to a group with the same exercise training but supplemented with placebo .This study is essentially exploratory in nature and designed to provide us with information to adequately develop power and execute a larger study. We have previously seen benefits from nitrate supplementation on function in PAD.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral Arterial Disease (ABI of less than 0.9)
* Diagnosed Type II Diabetes
* Intermittent Claudication for 3 or more months

Exclusion Criteria:

* Individuals with known alcohol or drug abuse problems
* Individuals who have suffered a heart attack or stroke, or have changes on a resting ECG, in the last 3 months
* Those classified as American Heart Association Class D
* Gangrene, impending limb loss or osteomyelitis
* Lower extremity vascular surgery, angioplasty or lumbar sympathectomy within 3 months of enrollment
* Severe peripheral neuropathy
* Any condition other than PAD that limits walking
* Chest pain during treadmill exercise which appears before the onset of claudication, or >3mm ST depression during exercise
* Subjects taking nitrates or nitroglycerin products
* Must not be taking protein pump inhibitor medications

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason D Allen, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Diet & Fitness Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Woessner M, VanBruggen MD, Pieper CF, Sloane R, Kraus WE, Gow AJ, Allen JD. Beet the Best? Circ Res. 2018 Aug 31;123(6):654-659. doi: 10.1161/CIRCRESAHA.118.313131. PMID 29976553
- See also: Frederick R. Cobb Non-Invasive Vascular Research Laboratory — http://cardiology.medicine.duke.edu/research/clinical-research/frederick-r-cobb-non-invasive-vascular-research-laboratory
- See also: Duke Clinical Trials Listing — http://www.dukehealth.org/clinicaltrials/20130131152500519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6,852 patients in Duke Cardiology and Vascular Surgery Clinics were screened, 392 potential study candidates were identified, and 18 subjects were enrolled from March 2013 through January 2014. Of the 18 subjects, 11 were randomized and 7 completed all study testing.
Period: Overall Study
Arm/Group | BR Juice (Beet-It Stamina Shot) & Supervised Exercise Training | BR Juice Placebo and Exercise Training
Started | 7 | 4
Completed | 5 | 2
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BR Juice (Beet-It Stamina Shot) & Supervised Exercise Training | BR Juice Placebo and Exercise Training | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (4.7) | 74.25 (5.1) | 71.63 (5.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Exercise Capacity - Maximal Oxygen Capacity (VO2peak)
Description: Exercise capacity will be assessed using a maximal cardiopulmonary exercise (CPX) test with expired gas analysis, for determination of peak oxygen consumption
Time Frame: Baseline & 16 Weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | BR Juice (Beet-It Stamina Shot) & Supervised Exercise Training | BR Juice Placebo and Exercise Training
Number analyzed (Participants) | 5 | 2
ml/kg/min | 0.85 (0.57) | -0.15 (1.13)

2. Primary Outcome: Change in Exercise Capacity - Time to Exhaustion (TTE)
Description: Exercise capacity will be assessed using a maximal cardiopulmonary exercise (CPX) test for determination of Time to Exhaustion (TTE)
Time Frame: Baseline & 16 Weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BR Juice (Beet-It Stamina Shot) & Supervised Exercise Training | BR Juice Placebo and Exercise Training
Number analyzed (Participants) | 5 | 2
seconds | 196.25 (201) | 247.5 (249.61)

3. Primary Outcome: Change in Exercise Capacity - Claudication Onset Time (COT)
Description: Exercise capacity will be assessed using a maximal cardiopulmonary exercise (CPX) test for determination of Claudication Onset Time (COT)
Time Frame: Baseline & 16 Weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BR Juice (Beet-It Stamina Shot) & Supervised Exercise Training | BR Juice Placebo and Exercise Training
Number analyzed (Participants) | 5 | 2
seconds | 189 (238.17) | 77.5 (36.06)

4. Secondary Outcome: Change in Functional Ability
Description: Six-Minute Walk test. This test simple and practical assessment of functional capacity. The test measures the distance that a patient can walk on a flat, hard surface in a period of 6 minutes. The test is self-paced and assesses the submaximal level of functional capacity. The subjects choose their own intensity and are allowed to stop and rest if necessary during the test.
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | BR Juice (Beet-It Stamina Shot) & Supervised Exercise Training | BR Juice Placebo and Exercise Training
Number analyzed (Participants) | 5 | 2
feet | 131 (288.08) | 47.5 (137.89)

5. Secondary Outcome: Change in Angiogenesis
Description: Gastrocnemious muscle biopsy will be performed to measure the number of capillaries per fibre as a marker of change in angiogenesis between groups.
Time Frame: Baseline and 16 weeks
Population: participants who underwent the gastrocnemius muscle biopsies
Measure: Mean (Standard Deviation); unit: ratio of capillaries to muscle fibres
Arm/Group | BR Juice (Beet-It Stamina Shot) & Supervised Exercise Training | BR Juice Placebo and Exercise Training
Number analyzed (Participants) | 2 | 0
ratio of capillaries to muscle fibres | 2 (0.22) |

6. Secondary Outcome: Change In Vascular Function
Description: Vascular Function will be measured as the Brachial artery flow-mediated dilation (BAFMD)
Time Frame: Baseline and 16 weeks
Population: participants who completed study
Measure: Number; unit: change % dilation
Arm/Group | BR Juice (Beet-It Stamina Shot) & Supervised Exercise Training | BR Juice Placebo and Exercise Training
Number analyzed (Participants) | 5 | 2
change % dilation | 1.83 | -3.56

ADVERSE EVENTS:
Arm/Group | BR Juice (Beet-It Stamina Shot) & Supervised Exercise Training | BR Juice Placebo and Exercise Training
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 0/7 | 0/4

LIMITATIONS AND CAVEATS:
The largest limitation to the study was the evolving knowledge on conversion rates of oral inorganic nitrate to nitrite. We found a good deal of unexpected inter and intra-subject variation in conversion rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes